CLINICAL TRIAL: NCT02381210
Title: Diagnosis and Prediction of Preeclampsia: A Case Control Study of the Clinical Utility of Congo Red Dot Test in Bangladesh and Mexico
Brief Title: Diagnosis and Prediction of Pre-Eclampsia by Using Congo Red Dot Test in Bangladesh and Mexico
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4004-A
Record Dates: First submitted 2015-02-25; First posted 2015-03-06 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2018-11

CONDITIONS: Preeclampsia
Keywords: Congo Red Dot Test
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CLINICALLY CONFIRMED PREECLAMPSIA: Pregnant women with clinical diagnosis of preeclampsia (severe, mild or superimposed) will provide a urine sample to determine the presence or absence of proteinuria using the Congo Red Dot test.
  Interventions: Device: Congo Red Dot Test
- CLINICALLY HEALTHY: Pregnant women admitted to the hospital for delivery of a healthy normal baby at term (induction of labor or an elective Caesarean Section) will provide a urine sample to determine the presence or absence of proteinuria using the Congo Red Dot test.
  Interventions: Device: Congo Red Dot Test

INTERVENTIONS:
Device: Congo Red Dot Test — The Congo Red Dot test is a simple test has been developed to detect unfolded or misfolded proteins in urine.

SUMMARY:
A cross sectional study design will evaluate the diagnostic value of the CRD test to the pregnant women attending the Dhaka Medical College Hospital and Hospital Materno-Infantil Inguarán, tertiary level facilities in Bangladesh and Mexico City.

DETAILED DESCRIPTION:
A cross sectional study design will evaluate the diagnostic value of the Congo Red Dot test to the pregnant women attending the Dhaka Medical College Hospital and Hospital Materno-Infantil Inguarán, tertiary level facilities in Bangladesh and Mexico City. Women attending the hospital with clinically confirmed cases of preeclampsia and clinically healthy women who deliver at term will be eligible for the study. Investigators will enroll about 200 women at each facility. Investigators will target the following women for enrollment: women with clinical diagnosis of preeclampsia (severe, mild or superimposed) (n=100); and clinically healthy women who deliver at term (n=100). The purpose of the research is to determine the clinical utility of congophilia (affinity for the dye Congo Red) in the diagnosis and prediction of preeclampsia. Investigators will determine the diagnostic value of this test by testing the urine sample provided to determine the presence or absence of proteinuria or congophilia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Willing to provide a urine sample
* Eligible to consent to research according to local laws and regulations
* Present with a clinical diagnosis of preeclampsia (severe, mild or superimposed) OR clinically healthy and delivering at term

Exclusion Criteria:

-None

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women attending Dhaka Medical College Hospital and Hospital Materno-Infantil Inguarán with clinically confirmed cases of preeclampsia and clinically healthy women who deliver at term will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of urine congophilia using Congo Red Dot test | within 1 month of urine sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Irina Buhimschi, Dr, Principal Investigator — Nationwide Children's Hospital; Beverly Winikoff, Dr, Principal Investigator — Gynuity Health Projects
Locations (2):
- Dhaka Medical College, Dhaka, Bangladesh
- Hospital Materno-Infantil Inguarán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided